CLINICAL TRIAL: NCT04421599
Title: Investigation of the Necessity of Aspiration During The Intramuscular Injection Administered in the Ventrogluteal Site and Its Effect on Pain
Brief Title: Necessity of Aspiration in the Ventrogluteal Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Leyla BARAN, Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000-0001-7881-8556
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Nursing; Injection Site
Keywords: Ventrogluteal area; aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A (Experimental): Experimental Group A who were administered intramuscular injection during which aspiration lasted for 5-10 seconds.
  Interventions: Other: The Necessity of Aspiration
- Control Group (No Intervention): Control Group who were administered intramuscular injection during which aspiration lasted for 1-2 seconds.
- Experimental Group B (Experimental): Experimental Group B who were not administered aspiration during IM injection.
  Interventions: Other: The Necessity of Aspiration

INTERVENTIONS:
Other: The Necessity of Aspiration — The patients who met the inclusion criteria and agreed to participate in the study were assigned to the Experimental Group A who were administered IM injection during which aspiration lasted for 5-10 seconds, to the Control Group who were administered IM injection during which aspiration lasted for 1-2 seconds, and to the Experimental Group B who were not administered IM injection according to the stratified block randomization list. The same "Intramuscular Injection Application Protocol" was applied while all the injections were administered.
  Arms: Experimental Group A; Experimental Group B

SUMMARY:
H1: Aspiration is not necessary for IM injections applied from the ventrogluteal region.

H2: Aspiration procedure increases pain in IM injections applied from ventrogluteal region.

H3: The duration of the aspiration procedure on IM injections applied from the ventrogluteal region is effective on pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient who came to the Emergency Service Care Unit for "Diclofenac Sodium" injection
* Have no vision and hearing problems,
* Who have no disease that may affect their perception of pain
* Who can evaluate the "Visual Analog Scale" correctly, scoring 5 points or less from the VAS,
* Body Mass Index is between 18.5-24.9 kg / m2,
* Who do not have any discomfort in the extremities that will prevent them from taking the desired position,
* No complications due to intramuscular injections such as abscess, infection, tissue necrosis and hematoma in the ventrogluteal region
* No nodules or masses in the area

Exclusion Criteria:

* Patients who refuse the injection are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 15 minutes
  The content of the study was explained to the patients coming to the emergency room. Written informed consents were obtained in line with the "Individual Introductory Information Form" of the patients.
  Individual Introductory Information Form: This form includes questions such as the patient's application group, diagnosis, age, gender, height, weight, and blood intake during aspiration in intramuscular injection. It is completed within the first 10-15 minutes of contact with the patient.
Visual Analog Scale (VAS) | 5 minutes
  Intramuscular injection was performed in accordance with the application group assigned to the patients who filled the Individual Introductory Information Form. The patients were not told which group they belonged to.
  A nurse who except the researcher who performed the application evaluated pain levels that patients feel during injection immediately after the intramuscular injection application, with a Visual Analog Scale. The minimum score that can be obtained from this scale is 0 and the maximum score is 10. A higher score indicates that the pain is more severe. This scale was applied in minutes 1-5 after intramuscular injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyea SC, Nicoll LH. Administration of medications via the intramuscular route: an integrative review of the literature and research-based protocol for the procedure. Appl Nurs Res. 1995 Feb;8(1):23-33. doi: 10.1016/s0897-1897(95)80279-7. PMID 7695353
- [Derived] Baran L, Gunes U, Donmez H. Investigation of the Necessity of Aspiration During the Intramuscular Injection Administered in the Ventrogluteal Site and Its Effect on Pain: A Randomized Controlled Trial. Clin Nurs Res. 2023 May;32(4):821-829. doi: 10.1177/10547738221136470. Epub 2022 Dec 20. PMID 36540016